CLINICAL TRIAL: NCT03534622
Title: A Phase I, Open-Label, Safety and Pharmacokinetic Study To Assess Bronchopulmonary Disposition of Intravenous Delafloxacin in Healthy Adults
Brief Title: Evaluate Safety and Pharmacokinetic To Assess Bronchopulmonary Disposition of Intravenous Delafloxacin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ML-3341-119
Record Dates: First submitted 2018-04-18; First posted 2018-05-23 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — delafloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Delafloxacin (Experimental): Dosing will be initiated on Day 1. All participants will receive 300-mg delafloxacin as a
  1-hour intravenous infusion every 12 hours (± 15 minutes) for a total of 7 doses.
  Interventions: Drug: Delafloxacin

INTERVENTIONS:
Drug: Delafloxacin — In this study, thirty subjects who meet the entry criteria will be assigned to 1 of 5 groups (A, B,C, D, or E) to receive 300 mg delafloxacin IV every 12 hours for a total of 7 doses over 4 days

SUMMARY:
The purpose of this study is to evaluate the steady-state intrapulmonary disposition of delafloxacin in healthy adult participants.

DETAILED DESCRIPTION:
This study will evaluate the safety and pharmacokinetics (PK) of delafloxacin in healthy adult participants by assessing the intrapulmonary disposition in adults receiving 300 mg delafloxacin IV every 12 hours for a total of 7 doses over 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant has no clinically important abnormal physical findings that could interfere with the conduct of the study.
* Participant has no clinically significant laboratory abnormalities.
* Participant has normal (or abnormal but not clinically significant) ECG measurements.
* Participant has BMI between 18.0 and ≤30.0 kg/m2, inclusive, or if outside the range, considered not clinically significant.
* Participant has normal (or abnormal but not clinically significant) blood pressure and pulse rate measurements. Blood pressure and pulse rate will be measured after the participant has been in a sitting position for 5 minutes. For this study, normal blood pressure is defined as 100 to 140 mmHg systolic and 50 to 90 mmHg diastolic, inclusive. Normal pulse rate is defined as 50 to 90 beats per minute, inclusive.
* Participant is willing and able to abstain from alcohol, caffeine, and methylxanthine containing beverages or food. Alcohol, caffeine, and methylxanthine consumption will be prohibited within 96 hours before Check-in and throughout the entire study throughout Follow-up.
* Participant is able to communicate well with the investigator and comply with the requirements of the entire study.
* Participant provides written informed consent to participate as indicated by a signature on the informed consent form (ICF).
* Participant agrees to use an adequate method of contraception during the study and for 30 days after the final dose. Female partners of male subjects should also use an additional reliable method of contraception. Adequate methods of contraception for the participant and partner include, but are not limited to, condoms with spermicide gel,diaphragm with spermicide gel, hormonal or nonhormonal intrauterine device, surgical sterilization, vasectomy, oral contraceptive pill, depot progesterone injections, or abstinence. If abstinence is indicated as the method of contraception, the participant must have been abstinent for 6 weeks before enrollment in the study. If a participant is usually not sexually active but becomes active, the participant and his or her partner should use one of the listed contraceptive methods.
* Female subjects of childbearing potential must be nonpregnant, nonlactating, and have a negative serum human chorionic gonadotropin pregnancy test at Screening and a negative urine pregnancy test at Check-In.

Exclusion Criteria:

* Participant has received any investigational drug within 30 days before administration of the first dose of the study drug (6 months for biologic therapies) or 5 half-lives of the investigational drug, if known, whichever time period is longer.
* Participant has received delafloxacin previously.
* Participant is a female who is pregnant or breastfeeding. Pregnancy status will be confirmed by serum assay for qualitative human chorionic gonadotropin at Screening and a urine assay performed at Check-in.
* Participant has a positive test result for alcohol, amphetamines, barbiturates, benzodiazepines, cocaine metabolites, opiates, cannabinoids, or cotinine, at Screening or Check-in.
* Participant has a positive screening test for hepatitis B surface antigen, hepatitis C antibody, and/or human immunodeficiency virus antibodies.
* Participant has any surgical or medical condition that, in the judgment of the investigator,might interfere with the absorption, distribution, metabolism, or excretion of the study drug.
* Participant has used any medication (prescription or over-the-counter [OTC], including health supplements and herbal remedies, with the exception of acetaminophen (as described in Exclusion Criterion 9) within 2 weeks (4 weeks for enzyme inducers including St John's wort [Hypericum perforatum]) or 5 half-lives (whichever is longer) before the first dose of study drug.
* Participant has used an oral or IV antibiotic within 3 months of administration of the first dose of the study drug.
* Participant has routinely or chronically used more than 1 g of acetaminophen daily.
* Participant has performed strenuous activity, sunbathing, and/or contact sports within 96 hours (4 days) before Check-in on Day -1. The participant should abstain from these activities for the duration of the study.
* Participant has donated or lost greater than 400 mL of blood in the 30 days before administration of the first dose of study drug.
* Participant is unable to be venipunctured or tolerate venous access as determined by the investigator or designee.
* Participant has a history of any significant drug allergy (such as anaphylaxis or hepatotoxicity) or drug reaction (angioedema, atopic dermatitis, or uticaria), including medical history of significant hypersensitivity or allergic reaction to quinolones or beta-lactam antibiotics, lidocaine, or similar compounds. Participants with a history of seasonal allergies are allowed unless the allergy is active or has required treatment within the past 30 days.
* Participant has a history of clinically significant, clinically relevant hematologic, renal, hepatic, bronchopulmonary (including history of chronic respiratory disorders, anatomy not conducive for bronchoscopy), neurological, psychiatric, metabolic, endocrine disorder (eg, diabetes, thyroid disease) or cardiovascular disease, in the opinion of the investigator.
* Subject has a history of clinically significant GI disease, or gastroenteritis (vomiting or diarrhea) or any history of GI bleeding (excluding bleeding from hemorrhoids), and/or surgery that would result in the subject's inability to absorb or metabolize the study drug (eg, gastrectomy, gastric bypass, cholecystectomy).
* Participant has a history of any drug or alcohol abuse in the past 2 years, or alcohol consumption greater than 21 units per week in males and 14 units per week in females. A unit of alcohol is equivalent to 1 can of beer, 1 glass of wine, or the equivalent of 1 alcoholic drink. Alcohol consumption will be prohibited within 96 hours before Check-in on Day -1 and throughout the entire study until Follow-up.
* Participant currently smokes or has smoked in the past year or uses or has used nicotine or nicotine containing products in the past 6 months.
* Participant has had any major surgery within 4 weeks of study drug administration.
* Participant has a history of malignancy within the past 5 years other than past history of localized or surgical removal of focal basal cell skin cancer, cervical cancer in situ treated successfully in the past by local treatment (including but not limited to cryotherapy or laser therapy), or by hysterectomy.
* Participant has any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participants in the study.
* Participation in another clinical study within 30 days of enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Delafloxacin plasma PK:Tmax | Day 4
Delafloxacin plasma PK: Cmax | Day 4
Delafloxacin plasma PK: AUCτ | Day 4
Delafloxacin plasma PK: AUC0-t | Day 4
Delafloxacin plasma PK: AUCinf | Day 4
Delafloxacin plasma PK: T1/2 | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Sue K Cammarata, MD, Study Director — CMO, MelintaTherapeutics, Inc.
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Horcajada JP, Salata RA, Alvarez-Sala R, Nitu FM, Lawrence L, Quintas M, Cheng CY, Cammarata S; DEFINE-CABP Study Group. A Phase 3 Study to Compare Delafloxacin With Moxifloxacin for the Treatment of Adults With Community-Acquired Bacterial Pneumonia (DEFINE-CABP). Open Forum Infect Dis. 2019 Dec 5;7(1):ofz514. doi: 10.1093/ofid/ofz514. eCollection 2020 Jan. PMID 31988972